CLINICAL TRIAL: NCT00052169
Title: A Phase 2, Multi-Center Trial of ZD1839 (IRESSA) in Combination With Docetaxel as First-Line Treatment in Patients With Advanced Breast Cancer
Brief Title: Therapy With Docetaxel and ZD1839 for Patients Who Have Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Norman Wolmark, MD/Chairman, NSABP Foundation Inc., NSABP Foundation, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FB-IR-002
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Breast Neoplasms
Keywords: metastatic breast cancer; docetaxel; Taxotere; ZD 1839; gefitinib; NSABP; advanced breast cancer; AstraZeneca
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ZD1839 in combination with docetaxel — Docetaxel given as 75 mg/m2 IV every 3 weeks combined with ZD1839 (IRESSA) 250 mg orally daily until disease progression or withdrawal criteria are met.
  Other Names: Docetaxel (Taxotere); ZD1839, gefitinib (Iressa)

SUMMARY:
The purpose of this study is to learn how breast cancer tumors respond to treatment combining the drugs docetaxel and ZD1839.

DETAILED DESCRIPTION:
Patients with advanced breast cancer continue to have an extremely poor prognosis with an average life expectancy of approximately 2 years. Novel treatments designed to exploit biologic properties of the tumor are urgently required as a means to improve the outcome for the large numbers of patients who relapse after receiving optimal chemotherapy treatments.

Overexpresssion of EGFR and/or TGF-alpha is frequent in human breast cancer and has been correlated in many cases with poor prognostic features. Inhibition of the EGFR pathway has been proposed as a potential therapeutic modality in advanced breast cancer. The antiproliferative activity of ZD 1839 in combination with cytotoxic drugs, such as docetaxel was evaluated in breast cancer cell lines ZR-75-1 and MCF-10A ras that coexpress EGFR and TGF-alpha. Combination treatment demonstrated dose dependent supra-additive growth inhibition and markedly enhanced apoptotic cell death.

Although taxanes bind to the microtubular network in cells that is essential for mitotic and interphase cellular functions, the mechanism by which these agents induce cell death is not entirely clear. Docetaxel has also shown dose-dependent anti-angiogenic activity. Thus, the mechanism(s) of anti-tumor activity of docetaxel remain unclear and combinations of signal transduction pathway inhibition and/or anti-angiogenesis may provide potentiation of concurrent ZD 1839 and docetaxel therapy.

This phase 2 trial is designed to prospectively investigate the efficacy and safetey of combination therapy with ZD 1839 and docetaxel in patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria

* Histologic confirmation of breast cancer
* Signed consent
* Current diagnosis of metastatic breast cancer
* At least one uni-dimensionally measurable lesion with clearly defined margins
* Patients taking bisphosphonates for documented prior bone metastasis may be included
* Patients may have received prior adjuvant chemotherapy including an anthracycline and/or an alkylating agent. Patients may have received prior paclitaxel or trastuzumab for adjuvant therapy. Patients may not have received prior docetaxel treatment
* Patients may have received unlimited prior hormonal therapy regimens for metastatic disease or adjuvant therapy and must have documentation of progressive disease prior to entry. Hormonal therapy must be discontinued at least 2 weeks prior to study entry
* Patients may have received prior radiation therapy provided it was completed at least 2 weeks before study entry. Prior radiotherapy to treat bone metastasis or spinal cord compression is permitted provided it was completed prior to study entry
* Zubrod performance status 0, 1, or 2
* Life expectancy of 12 weeks or more in opinion of investigator
* LVEF greater than or equal to LLN without clinical signs or symptoms of heart failure
* adequate bone marrow, hepatic, and renal function

Ineligibility Criteria

* Prior ZD1839 or other anti EGFR or small molecule TKI
* Previous or concurrent chemo or Herceptin for metastatic breast cancer
* Unresolved non-permanent major end organ chronic toxicity from previous anticancer therapy greater than CTC grade 2
* Radiation therapy less than 14 days before study entry, with exception of RT to treat bone metastasis or spinal cord compression
* Incomplete healing of surgical incision from previous major surgery
* Newly diagnosed (within 12 weeks) intracerebral metastases
* Signs of neurological symptoms consistent with new onset spinal cord compression
* Evidence of severe or uncontrolled systemic disease
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for patient to participate
* Pregnancy or breast feeding
* Patients who are currently using contact lenses. Patients who discontinue wearing contact lenses prior to study entry are eligible.
* Patients with untreated ocular inflammation or infection
* Patients with contraindications to corticosteroid use
* History of another malignancy within past 5 years that could confound diagnosis or staging of breast cancer
* Patients receiving other investigational drugs
* Previous docetaxel treatment
* Patients currently taking systemic retinoids or herbal medicines
* Patients currently taking drugs known to induce Cyt P4503A4

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To estimate the clinical benefit rate of the combination of ZD 1839 and docetaxel; clinical benefit measured by clinical response, pathologic response, and stable disease (SD greater than or equal to 24 weeks) | 2 years
To characterize the safety profile of the combination of ZD 1839 and docetaxel as measured by the frequency and severity of adverse events. | 2 years

SECONDARY OUTCOMES:
To estimate the duration of clinical benefit. | 2 years
To estimate the objective tumor response rate (using RECIST best overall response of CR + PR). | 2 years
To estimate the duration of tumor response. | 2 years
To estimate progression-free survival. | 2 years
To estimate time to treatment failure by measuring time to treatment failure (includes disease progression, second primary cancer, death from any cause, or discontinuation of protocol therapy in the absence of disease progression). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (1):
- NSABP Operations Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Dennison SK, Jacobs SA, Wilson JW, Seeger J, Cescon TP, Raymond JM, Geyer CE, Wolmark N, Swain SM. A phase II clinical trial of ZD1839 (Iressa) in combination with docetaxel as first-line treatment in patients with advanced breast cancer. Invest New Drugs. 2007 Dec;25(6):545-51. doi: 10.1007/s10637-007-9055-6. Epub 2007 Jun 12. PMID 17563856